CLINICAL TRIAL: NCT02356640
Title: A Randomized Controlled Trial on Endoscopic Ultrasound-guided Celiac Ganglion Neurolysis Versus Percutaneous Celiac Plexus Neurolysis in Patients With Inoperable Cancer
Brief Title: EUS-guided CGN for Inoperable Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EUSCGN-02
Record Dates: First submitted 2014-08-20; First posted 2015-02-05 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Intractable Abdominal Pain Secondary to Inoperable Malignancy
Keywords: Celiac plexus neurolysis; Celiac ganglion neurolysis; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-guided celiac ganglion neurolysis (Active Comparator): Endoscopic ultrasound guided celiac ganglion neurolysis would be performed
  Interventions: Procedure: EUS-guided celiac ganglion neurolysis; Device: Olympus UM 2000
- Percutaneous celiac plexus neurolysis (Active Comparator): Percutaneous celiac plexus neurolysis would be performed
  Interventions: Procedure: Percutaneous celiac plexus neurolysis; Device: B-D Quincke Type Point; Drug: Levobupivacaine

INTERVENTIONS:
Procedure: EUS-guided celiac ganglion neurolysis — EUS-CGN would be performed with a linear video echoendoscope (Olympus UM 2000; Olympus Co Ltd, Japan). The celiac ganglia are visualized under linear EUS and the injection would be applied directly into the ganglia. It is represented by small 2 to 3 mm hypoechoic nodules with hyperechoic foci in the center or a single elongated hypoechoic structure. IIf the ganglia are not identified by EUS, then injection would be performed as bilateral injections at the celiac vessel trunk. All procedures would be performed by a two experienced endosonographer.
  Arms: EUS-guided celiac ganglion neurolysis
Procedure: Percutaneous celiac plexus neurolysis — Percutaneous fluoroscopy-guided CPN would be performed in the operation theatre with the transcural technique. A 22-gauge, 17 cm-long spinal needle (B-D Quincke Type Point, Becton Dickinson &Co., NJ 07417, USA) would be inserted and advanced just caudal to the margin of 12th rib and cephalad to the transverse process of L1 toward the anterolateral surface of the L1 vertebral body. Final needle position would be confirmed by radiographic contrast, layering over anterior surface of aorta. 10mL of levobupivacaine (0.25%), followed by 10mL of absolute alcohol would be injected on both sides using separate punctures.
  Arms: Percutaneous celiac plexus neurolysis
Device: Olympus UM 2000
  Arms: EUS-guided celiac ganglion neurolysis
Device: B-D Quincke Type Point
  Arms: Percutaneous celiac plexus neurolysis
Drug: Levobupivacaine
  Arms: Percutaneous celiac plexus neurolysis

SUMMARY:
Patients suffering from pancreatic cancer are associated with a poor prognosis and survival of less than one year is expected in inoperable tumours. Management of these patients would be towards palliation of symptoms. Severe pain occurs in 50 to 70% of the patients and this "intractable" pain is often difficult to treat. Different pharmacological agents have been used in the past to control this pain and these include non-steroidal anti-inflammatory drugs and narcotic agents. However, patients' responses are often variable and difficult to predict. Furthermore, these agents are associated with their own adverse effects and may further impair quality of life.

Celiac plexus neurolysis (CPN) was first described in 1919, since then, different approaches of performing the procedure have been described. The standard technique involves a percutaneous approach but CPN can also be performed by an intra-operative approach with open or laparoscopic means. Results from meta-analysis have shown that CPN was associated with superior pain relief as compared to analgesic therapy alone and reduces the need for opioids analgesics in patients with inoperable pancreatic cancer. Furthermore, CPN causes fewer adverse effects than opioid analgesics and it is the preferred method of improving pain relief in these patients.

Recently, endoscopic ultrasonography (EUS) - guided CPN has become popular. The approach is safe and effective and was shown to be associated with long lasting pain relieve in patients suffering from chronic pancreatitis or pancreatic cancer. Serious complications are uncommon and are less than 2% in these series. Transient diarrhoea and hypotension are common after CPN and is seen up to 30% to 40% of the patients, regardless of whether the procedure is being done by the EUS or percutaneous approach. The EUS approach offers several theoretical advantages over the percutaneous option. Most notably is the visualization of the celiac ganglia situated anterior to the aorta, allowing direct injection of the ganglia with alcohol resulting in celiac ganglion neurolysis (CGN). This increases the accuracy of CPN and may result in improved pain control. Furthermore, it could reduce complications associated with the percutaneous approach that includes lower extremity paresthesia and paralysis.

Hence, the aim of the study is to compare the efficacy and safety of endoscopic ultrasound (EUS)-guided celiac ganglion neurolysis (CGN) versus percutaneous celiac plexus neurolysis (CPN) in reducing cancer pain in patients suffering from inoperable cancer. With direct visualization and injection of the celiac ganglion, the investigators hypothesis that EUS-guided CGN is more advantageous on improving pain relief and decreasing the need for opioid analgesics in patients with inoperable cancer as compared to percutaneous CPN.

ELIGIBILITY:
Inclusion Criteria:

1. All patients ≥ 18 years old with cytology or histology confirmed pancreatic cancer, or radiologically suggestive of pancreatic cancer ( for patients whom biopsy is impossible)
2. Pain associated with inoperable cancer ( including abdominal pain or back pain, managed according to WHO analgesic ladder, with VAS score ≥4 despite simple analgesics (first 2 steps of WHO analgesic ladder)
3. Inoperability of cancer as demonstrated by EUS, computed tomography (CT) or Positive emission tomography
4. Informed consent available

Exclusion Criteria:

1. Unable to safely undergo EUS for any reason
2. Patient is unable to lie prone for procedure
3. Coagulopathy (prolongation of prothrombin time > 18 sec) or thrombocytopenia <80,000 platelets/ml)
4. Previous CPN or other neurolytic block that could affect pancreatic cancer-related pain or had implanted epidural or intrathecal analgesic therapy
5. Another cause for abdominal pain such as pseudocyst, ulcer or other intra-abdominal disorder
6. Allergy to local anaesthesia, contrast, or alcohol
7. Potential patient noncompliance (refusing to follow schedule of events)
8. Active alcohol or other drug use or significant psychiatric illness
9. Expected survival less than 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-08; Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Pain score measured using the visual analogue scale | 2 weeks
  Pain scores at 2 weeks after the procedure will be measured using the visual analogue scale

SECONDARY OUTCOMES:
Opioid requirements (Amounts of opioid medications required at assessment interval) | 2 weeks then monthly for 1 yr or till death
  Amounts of opioid medications required at assessment interval
Adverse events | 2 weeks, then monthly for 1 yr or till death
  Patients would be monitored for presence of adverse events after CGN or CPN. Transient diarrhea and hypotension are common manifestations of the sympathetic blockade and may be seen in up to 38 and 44 percent of the patients. Severe adverse effects after percutaneous CPN include neurologic complications (l%) such as lower extremity weakness and paresthesia, epidural anesthesia, and lumbar puncture. Non-neurological adverse effects (1%) including pneumothorax, shoulder, chest and pleuritic pain, hiccoughing, and hematuria have also been reported.
Quality of life scores (FACT-Hep Chinese module) | 2 week, then monthly for 1 yr or till death
  QOL would be assessed using the FACT-Hep Chinese module

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Wyse JM, Carone M, Paquin SC, Usatii M, Sahai AV. Randomized, double-blind, controlled trial of early endoscopic ultrasound-guided celiac plexus neurolysis to prevent pain progression in patients with newly diagnosed, painful, inoperable pancreatic cancer. J Clin Oncol. 2011 Sep 10;29(26):3541-6. doi: 10.1200/JCO.2010.32.2750. Epub 2011 Aug 15. PMID 21844506
- [Background] Levy MJ, Topazian MD, Wiersema MJ, Clain JE, Rajan E, Wang KK, de la Mora JG, Gleeson FC, Pearson RK, Pelaez MC, Petersen BT, Vege SS, Chari ST. Initial evaluation of the efficacy and safety of endoscopic ultrasound-guided direct Ganglia neurolysis and block. Am J Gastroenterol. 2008 Jan;103(1):98-103. doi: 10.1111/j.1572-0241.2007.01607.x. Epub 2007 Oct 26. PMID 17970834
- [Background] Doi S, Yasuda I, Kawakami H, Hayashi T, Hisai H, Irisawa A, Mukai T, Katanuma A, Kubota K, Ohnishi T, Ryozawa S, Hara K, Itoi T, Hanada K, Yamao K. Endoscopic ultrasound-guided celiac ganglia neurolysis vs. celiac plexus neurolysis: a randomized multicenter trial. Endoscopy. 2013;45(5):362-9. doi: 10.1055/s-0032-1326225. Epub 2013 Apr 24. PMID 23616126